CLINICAL TRIAL: NCT03642171
Title: A Post Market Surveillance Study of the Performance and Safety of UT 380® Contraceptive Intra Uterine Device in Nulliparous, Uniparous and Multiparous Women
Brief Title: Surveillance Study of the Contraceptive Intrauterine Device UT380®
Acronym: CCDDIUUT
Status: Completed | Type: Observational
Sponsor: Quanta Medical (Industry)
Collaborators: Prodimed S.A. (Other); CCD (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2868
Record Dates: First submitted 2018-07-16; First posted 2018-08-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-03

CONDITIONS: Contraceptive; Complications, Intrauterine
Keywords: Contraception; Intrauterine Device; UT380

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is a long term Post Market Surveillance Study involving women who will received UT 380® device as a contraceptive method.

DETAILED DESCRIPTION:
Prospective data on contraceptive performance of the UT380® from a large number of women are not yet available. Here we describe a long term Post Market Surveillance Study involving women who will received UT 380® device as a contraceptive method. Reports of case series usually contain detailed information about the individual patients. This includes demographic information (e.g. age and gender) and information on diagnosis, treatment, response to treatment, follow-up after treatment and patients experience of the treatment. In addition, it also include the health care staff's experience of the use of the UT 380. The result of this study will be used for different purposes e.g. marketing activities such as posters, folders, or targeted journals and/or conferences.

ELIGIBILITY:
Inclusion Criteria:

* Woman > 18 years old
* nulliparous, uniparous and multiparous
* not currently using a contraceptive method or are willing to switch to a new reversible contraceptive
* with an indication of implantation of a UT380® IUD
* agreeing to participate in the study

Exclusion Criteria:

* Patient with risk of post implantation bleeding or high level of bleeding during menstruation period
* Patient with a risk of infection
* Patient that meet any of the absolute contraindication of UT 380®
* Any other elements that the investigator may think relevant and cannot allow the use of UT380®

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — UT380® is intended to be used in nulliparous, uniparous and multiparous women
Study Population: The patients will be recruited in France city privates practicing gynaecologist.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Unintended pregnancy rate | 5 years
  Unintended pregnancy rate
Device expulsion rate | 5 years
  Device expulsion rate
Discontinuation rate | 5 years
  Discontinuation rate

SECONDARY OUTCOMES:
Extra uterine pregnancy rate | 5 years
  Extra uterine pregnancy rate
Assessment of physicians satisfaction regarding the use of the UT380 using 5 points likert scale (1: not at all satisfied 5: very satisfied) | 5 years
  Physicians satisfaction regarding the use of the UT 380 will be assessed at post implantation visit (2 visits the fisrt year, and one visit per years during the following 4 years) using 5 points likert scale (1: not at all satisfied 5: very satisfied)
Assessment of patients satisfaction regarding the use of the UT 380® using 5 points likert scale (1: not at all satisfied 5: very satisfied) | 5 years
  Patients satisfaction regarding the use of the UT 380® will be assessed at post implantation visit (2 visits the fisrt year, and one visit per years during the following 4 years) using 5 points likert scale (1: not at all satisfied 5: very satisfied)
Removal rate of the UT380® due to excessive bleeding | 5 years
Removal rate of the UT380® due to pain | 5 years
Removal rate of the UT380® due to pelvic inflammatory diseases | 5 years
Removal rate of the UT380® due to other disease relevant in the contexte of the trial | 5 years
Removal rate of the UT380® due to desired pregnancy | 5 years
Removal rate of the UT380® due to any other personal reason | 5 years
Removal rate of the UT380® due to investigator decision | 5 years
Safety data such as uterin perforation | 5 years
  Uterin perforation rate
Safety data such as any issue occurring immediately after the implantation of the device | 5 years
  Rate of issue occurring immediately after the implantation of the device
Safety data such as any issue occurring between two visits: Abdominopelvic or uterine pain outside the menstrual cycle, bleeding, | 5 years
  Rate of issue occurring between two visits
Safety data such as any issue during the device removal (such as pain, breaking device, excessive pulling force…) | 5 years
  Rate of issue during the device removal

CONTACTS AND LOCATIONS:
Locations (1):
- Quanta Medical, Boulogne-Billancourt, France